CLINICAL TRIAL: NCT02180009
Title: Dynamic Changes of Tim-3 on Monocytes and Soluble Tim-3 in Patients With Sepsis
Status: Completed | Type: Observational
Sponsor: Chinese PLA General Hospital (Other)
Collaborators: Beijing Institute of Basic Medical Science (Other)
Responsible Party: Principal Investigator, Feifei Ren, doctor of Department of Respiratory Medicine, Chinese PLA General Hospital
Other Study IDs: ZS2012009
Record Dates: First submitted 2014-07-01; First posted 2014-07-02 (Estimated); Last update posted 2016-01-28 (Estimated); Status verified 2016-01

CONDITIONS: Sepsis; Severe Sepsis; Septic Shock
MeSH Terms: conditions — Sepsis; Shock, Septic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples With DNA — peripheral blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- normal control: healthy people
- sepsis: mild response to infection
- severe sepsis: infection with at least one organ dysfunction
- septic shock: patients with septic shock

SUMMARY:
In this study, the investigators will dynamically detect the expression of an immune regulator- T cell Ig and mucin domain protein 3 (Tim-3) in patient with sepsis.

DETAILED DESCRIPTION:
In this study, we will collect the peripheral blood of 1,3,5,7,10,14 day after diagnose of sepsis.All the patients rolled in this study will be divided into three groups which is sepsis, severe sepsis and septic shock group according their severity. Then,the flow cytometry will be used to detect the express of Tim-3 on monocyte and ELISA will be used to exam the plasm soluble Tim-3.IL-6,IL-10,IL-12 and TNF-αin the peripheral blood will also be detected. We would like to find a new marker to predict the severity and prognosis of sepsis patients.

ELIGIBILITY:
Inclusion Criteria:

* More than one of the following:

clinical manifestations: (1) a body temperature greater than 38℃ or less than 36℃; (2) a heart rate greater than 90 beats/minute; (3)tachypnea, manifested by a respiratory rate greater than 20 breaths per minute, or hyperventilation, as indicated by a PaCO2 of less than 32 mmHg; and (4)an alteration in the white blood cell count, such as a count greater than 12×10^9/L, a count less than 4×10^9/L, or the presence of more than 10 percent immature neutrophils

Exclusion Criteria:

* (1)patients younger than 18 years of age; (2)agranulocytosis (granulocyte counts,0.5×10^9/L); (3) those discharged within 24 h; (4) those diagnosed with HIV infection or cancer; and (5) patients who refused to participate.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients with sepsis
Sampling Method: Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2013-12; Primary Completion 2015-08 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
all cause mortality | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Lixin Xie, PhD & MD, Principal Investigator — Head of Department of Respiratory Medicine,Chinese PLA Gerneral Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] Levy MM, Fink MP, Marshall JC, Abraham E, Angus D, Cook D, Cohen J, Opal SM, Vincent JL, Ramsay G; International Sepsis Definitions Conference. 2001 SCCM/ESICM/ACCP/ATS/SIS International Sepsis Definitions Conference. Intensive Care Med. 2003 Apr;29(4):530-8. doi: 10.1007/s00134-003-1662-x. Epub 2003 Mar 28. PMID 12664219